CLINICAL TRIAL: NCT01699230
Title: Potential Effects of Omega 3 Supplementation on Cardiomyocytes Membranes for Patients With Coronary Atherosclerosis?
Acronym: CORONOMEGA3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CHU-0120
Record Dates: First submitted 2012-07-13; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Atherosclerosis
Keywords: Elective cardiac surgery; with sternotomy and; cardiopulmonary bypass; for coronary artery; bypass graft.
MeSH Terms: conditions — Coronary Artery Disease | interventions — Docosahexaenoic Acids

ARMS (2):
- Omega 3 supplemented patients (Experimental): To show the existence of a atrial cardiomyocytes membranes modification in omega-3 supplemented patients with coronary atherosclerosis
  Interventions: Dietary Supplement: Omega 3
- Control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Omega 3 — To show the existence of a atrial cardiomyocytes membranes modification in omega-3 supplemented patients with coronary atherosclerosis
  Arms: Omega 3 supplemented patients

SUMMARY:
To show the existence of a atrial cardiomyocytes membranes modification in omega-3 supplemented patients with coronary atherosclerosis.

DETAILED DESCRIPTION:
Very few human data are currently available on the fatty acid composition of cardiomyocytes membranes. Preoperative omega-3 supplementation for patients undergoing cardiac surgery with cardiopulmonary bypass is correlated with a decreased frequency of postoperative complications in type of arrhythmia atrial fibrillation. Atrial fibrillation is the most common complication: 30 to 50% after myocardial revascularization. The occurrence of atrial fibrillation increases morbidity and mortality after surgery for sure. The pathophysiological mechanisms of common atrial fibrillation treated in heart rhythm units are different from those of postoperative atrial fibrillation. Indeed, atrial fibrillation is a common disease primarily of the left atrium, although atrial fibrillation after cardiac surgery is a multifactorial disease with implication of various pathogens such as inflammation without precise anatomical support. The preventive use of polyunsaturated fatty acids omega-3 long-chain (LC-AGPIω3), prior cardiac surgery is far from widespread due to a Lack of information dissemination, by insufficient number of published studies, despite the existence of a number of ongoing clinical trials and a complete ignorance of biological mechanisms of action. A human clinical study is needed. In a context of cardiac surgery with cardiopulmonary bypass and without deleterious side effects of preoperative enrichment in omega-3, it seems appropriate to conduct a feasibility study to provide information on structural changes in membranes of cardiomyocytes.

ELIGIBILITY:
Inclusion Criteria:

* Men without diabetes,
* over 50 years with overweight (BMI greater than 25) and
* without severe obesity (BMI less than 40)
* Patients who have given their written consent,
* the beneficiary of a social security system.
* Elective cardiac surgery with sternotomy and cardiopulmonary bypass for coronary artery bypass graft.

Exclusion Criteria:

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
fatty acid variations | at J-21

SECONDARY OUTCOMES:
postoperative arrhythmias (atrial fibrillation) | at J-21, J0, J7 and J30
postoperative inflammatory syndrome | at J-21, J0, J7 and J30

CONTACTS AND LOCATIONS:
Overall Officials: Kasra AZARNOUSH, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France